CLINICAL TRIAL: NCT07046637
Title: Short-Term Effects of Inspiratory Muscle Warm-Up and Fatigue on Diaphragmatic Function in Professional Basketball Players: A Randomized Controlled Trial
Brief Title: Acute Effects of Inspiratory Muscle Load on Diaphragmatic Recovery in Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 020
Record Dates: First submitted 2025-06-29; First posted 2025-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Sports Physical Therapy; Athletic Injuries; Healthy
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle fatigue group (Experimental): The EG (experimental group) will perform the diaphragmatic fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their MIP (Maximum Inspiratory Pressure) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.
  Interventions: Device: Inspiratory muscle fatigue group
- Inspiratory muscle warm-up group (Active Comparator): The inspiratory muscle warm-up group will perform the protocol of 2 sets of 30 repetitions at 40% of their MIP, one-on-one, and in a single session, breathing against submaximal inspiratory loads using a threshold valve device. The participants will follow a free pattern of breathing until complete the protocol.
  Interventions: Device: Inspiratory muscle warm-up group

INTERVENTIONS:
Device: Inspiratory muscle fatigue group — The subjects will perform deep inspirations against a threshold device with varying resistances
  Other Names: Inspiratory muscle fatigue
  Arms: Inspiratory muscle fatigue group
Device: Inspiratory muscle warm-up group — The subjects will perform deep inspirations against a threshold device with varying resistances
  Other Names: Inspiratory muscle warm-up
  Arms: Inspiratory muscle warm-up group

SUMMARY:
This randomized controlled trial investigates the acute effects of inspiratory muscle warm-up and fatigue on diaphragmatic function in professional basketball players. Using ultrasound imaging and maximal inspiratory pressure (PIM) assessment, the study evaluates changes in diaphragmatic thickness and respiratory strength before and after specific inspiratory muscle loading protocols. Findings aim to clarify the short-term impact of these interventions on diaphragmatic recovery capacity, with potential implications for respiratory training, performance enhancement, and injury prevention strategies in elite athletic populations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female professional basketball players aged between 18 and 35 years.
* Holding a valid federation license at the autonomous or higher competitive level.
* A minimum of 3 consecutive seasons of competition in official FEB, FIBA, or equivalent regional leagues.
* Regular training frequency of ≥4 sessions per week over the past 6 months.
* No previous experience with inspiratory muscle training.
* Ability to understand study procedures and provide written informed consent.

Exclusion Criteria:

* History of chronic respiratory, neuromuscular, or cardiovascular disease.
* Musculoskeletal injury limiting inspiratory effort or physical participation (current or within the past three months).
* Previous thoracic or abdominal surgery.
* Current smokers.
* Use of pharmacological treatments that could affect respiratory or muscular function.
* Participation in another interventional study within the past 4 weeks.
* Inability to understand or follow study instructions.
* Tympanic membrane perforation or middle/inner ear pathology.
* Pregnancy or postpartum period within the last 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | Immediately before intervention, immediately after intervention, 15 minutes post intervention and 30 minutes post intervention
  It will be assessed using a Breathare MIP/MEP® (GH Innotek Co., Ltd., Busan, Republic of Korea).The Breathare MIP/MEP® is likely a respiratory pressure meter or manometer designed for measuring respiratory muscle strength. It typically includes a mouthpiece connected to a pressure sensor, and the device measures the force or pressure generated during respiratory maneuvers.
  The person will be instructed to take a maximal deep breath in, and then exhale to residual volume. After that, they will be asked to inhale forcefully against the resistance provided by the Breathare MIP/MEP®. This measures the strength of the inspiratory muscles.
  The measures will be expressed in cmH2O.

SECONDARY OUTCOMES:
Diaphragmatic thickness and thickening fraction | Immediately before intervention, immediately after intervention, 15 minutes post intervention and 30 minutes post intervention
  The linear array probe with a frequency of 3.0-10 megahertz (MHz) is placed perpendicularly to chest wall close to the mid-axillary line which is between the 8th and 10th intercostal space. The thickness of diaphragm is measured at the end of expiration and maximum inspiration for three times and the average values were recorded.
  The measures will be expressed in centimeters.

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality and privacy considerations, individual participant data (IPD) will not be publicly available. However, de-identified data can be made available upon reasonable request to the corresponding author, subject to approval and adherence to ethical guidelines. The anonymity of participants will always be strictly maintained.

REFERENCES:
- [Derived] Ladrinan-Maestro A, Sanchez-Infante J, Rodriguez-Sanz D, Sanchez-Sierra A. Short-term effects of inspiratory muscle warm-up and fatigue on diaphragmatic function in professional basketball players: a randomized clinical trial. Eur J Appl Physiol. 2026 Jan 6. doi: 10.1007/s00421-025-06116-2. Online ahead of print. PMID 41493585